CLINICAL TRIAL: NCT00225108
Title: The Cesarean Section Thromboprophylaxis Pilot Study:A Randomized Open-Label Controlled Pilot Study of Prophylactic Low Molecular Weight Heparin in High Risk Postpartum Women Following Cesarean Section
Brief Title: The STOP CLOT Pilot Study: Study of Low Molecular Weight Heparin in High Risk Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2002191-01H
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; bleeding
MeSH Terms: conditions — Venous Thrombosis; Hemorrhage | interventions — Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin

SUMMARY:
Venous thromboembolism (VTE) remains the most common cause of maternal death in the developed world. VTE includes two conditions, deep vein thrombosis (DVT) and pulmonary embolism (PE). DVT refers to a blood clot that has formed in a deep vein, often in the legs and/or pelvis and PE refers to the passage of these clots into the lungs (which can be fatal). VTE is up to 10 times more common in pregnant women than non-pregnant women of comparable age. More than a third of pregnancy related VTE occur during the 6 weeks after delivery. When compared with vaginal delivery, cesarean delivery further increases the risk of pregnancy associated VTE by three-fold.

A medication called low molecular weight heparin is sometimes prescribed during pregnancy and after delivery to prevent VTE. However, clinical practice varies because there hasn't been adequate research to determine that this medication is safe and effective at preventing VTE during this time. The potential benefits of the medication must also be weighed against its cost and possible side effects.

The researchers are conducting a study that will assess the effectiveness and safety of low molecular weight heparin in women who are at moderate to high risk of VTE after a cesarean section. They will monitor these women to determine if those who received the medication have fewer blood clots. Participants will also be monitored closely for any side effects.

DETAILED DESCRIPTION:
BACKGROUND: Venous thromboembolism (VTE) remains the most common cause of maternal mortality in the developed world. VTE is up to 10 times more common in pregnant women than non-pregnant women of comparable age. More than a third of pregnancy related VTE occur during the brief postpartum period (6 weeks). When compared with vaginal delivery, cesarean delivery further increases the risk of pregnancy associated VTE by three-fold. Pregnancy associated VTE is unique in that isolated iliac vein thrombosis is more likely and long term morbidity (post-phlebitic syndrome) is common.

There is an absence of randomized controlled trials (RCTs) of thromboprophylaxis after C-section to guide practice. Many national societies have guidelines on thromboprophylaxis however these are not evidence based and compliance with these guidelines is poor. Thromboprophylaxis may be associated with adverse effects (bleeding, heparin induced thrombocytopenia, skin reactions), inconvenience and cost. It is critical that the efficacy and safety of thromboprophylaxis following cesarean delivery be assessed in well designed and conducted randomized trials.

OBJECTIVES: We are conducting a randomized double-blind placebo-controlled pilot study. The pilot study seeks to answer the question: Is a randomized double-blind placebo-controlled multicentre trial of low molecular weight heparin thromboprophylaxis feasible in moderate to high risk women post cesarean section with DVT detected by pelvic vein (MRV) or leg vein (leg compression ultrasound) imaging? Our ultimate goal is to determine:

1. Is LMWH effective in preventing postpartum DVT following cesarean section in women at moderate to high risk of VTE?
2. Is LMWH safe in preventing postpartum DVT following cesarean section in women at moderate to high risk of VTE?
3. Is LMWH cost effective in preventing postpartum DVT following cesarean section in women at moderate to high risk of VTE?

STUDY DESIGN: We propose a randomized double-blind placebo-controlled pilot study of prophylactic LMWH in women at moderate to high risk for VTE following cesarean section. Eligible, consenting and randomized participants will receive once-daily injections of study drug (4,500 IU tinzaparin sodium (Innohep®;) or placebo) within 6 to 24 hours postpartum and continue until 3 to 7 days postpartum. On the day of hospital discharge, bilateral leg imaging with compression leg ultrasounds and pelvic vein imaging with MRV will be completed. The primary outcome will be adjudicated DVT documented on ultrasounds or MRV on the day of hospital discharge. Secondary outcomes will include symptomatic DVT and PE, death from PE, major and minor bleeding, HIT during the six week postpartum period. All outcomes will be adjudicated by an independent committee of experts blinded to study drug allocation.

With a sample size of 134 patients we will have over 80% power to detect a 50% relative risk reduction in the primary outcome event rate and a large enough sample to determine the feasibility objectives of the pilot study (i.e. obtain a precise estimate of the primary outcome event rate [DVT], a precise estimate of the multicentre recruitment rate, feasibility and acceptability of blinded study drug and placebo administration, feasibility of obtaining local study centre MRV and central interpretation of MRV and a preliminary relative risk reduction estimate with study drug compared to placebo to inform final study sample size determination).

RELEVANCE: Maternal mortality is a devastating outcome with far reaching emotional and societal implications. Evidence to guide thromboprophylaxis in women at risk for the number 1 cause of maternal mortality is required.

ELIGIBILITY:
Inclusion Criteria (must meet inclusion criteria 1, 2 and 3):

1. At high risk for thromboembolism (any one of the following):

   1. Age > 35 years
   2. Obesity (> 80 kg)
   3. Para 4
   4. Gross varicose veins
   5. Current infection
   6. Pre-eclampsia
   7. Immobility prior to surgery (> 4 days)
   8. Major current disease: includes heart or lung disease, cancer, inflammatory bowel disease, and nephrotic syndrome.
   9. Emergency cesarean section in labour
   10. Extended major pelvic or abdominal surgery (e.g. cesarean hysterectomy)
   11. Patients with a family history of VTE
   12. History of superficial phlebitis
2. Delivered by cesarean section (emergency or planned)
3. Signed, informed consent

Exclusion Criteria (must not meet any of the following criteria):

1. Greater than 36 hours since delivery
2. Need for anticoagulation, including:

   1. Women with a confirmed thrombophilia
   2. Women with paralysis of lower limbs
   3. Women with personal history of VTE
   4. Women with antiphospholipid antibody syndrome (APLA)
   5. Women with mechanical heart valves
3. Contraindication to heparin therapy, including:

   1. History of heparin induced thrombocytopenia
   2. Platelet count of less than 100,000 x 10^6/L
   3. Hemoglobin <= 90 g/L or a greater than 30 g/L drop in hemoglobin compared to last antepartum result
   4. History of osteoporosis
   5. History of steroid use (one week or more)
   6. Active bleeding
   7. Documented peptic ulcer within 6 weeks
   8. Heparin, bisulfite, or fish allergy
   9. Severe hypertension (systolic blood pressure [SBP] > 200 and/or diastolic blood pressure [DBP] > 120)
   10. Severe hepatic failure (International Normalized Ratio [INR] > 1.8)
   11. Women with serum creatinine > 80 and an abnormal 24 hour creatinine clearance.
4. Contraindications to magnetic resonance imaging (MRI), including:

   1. Women with electrically, magnetically or mechanically activated implants
   2. Women with claustrophobia
5. Women < 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2006-09

PRIMARY OUTCOMES:
VTE on magnetic resonance venography (MRV) or bilateral leg Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Rodger MA, Avruch LI, Howley HE, Olivier A, Walker MC. Pelvic magnetic resonance venography reveals high rate of pelvic vein thrombosis after cesarean section. Am J Obstet Gynecol. 2006 Feb;194(2):436-7. doi: 10.1016/j.ajog.2005.07.044. PMID 16458642
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986